CLINICAL TRIAL: NCT05578846
Title: A Phase 1 Study to Assess the Bioequivalence Between 180 mg and 60 mg ALXN2050 Tablets and the Effect of Food on ALXN2050 Pharmacokinetics in Healthy Adult Participants
Brief Title: Bioequivalence Between 180 mg and 60 mg ALXN2050 Tablets and Food Effect on ALXN2050 Pharmacokinetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: ALXN2050-HV-112
Record Dates: First submitted 2022-10-11; First posted 2022-10-13 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Healthy Adult Participants
Keywords: Bioequivalence; Effect of Food

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Treatment sequence ABC (Experimental): Participants will be administered Treatment A (3 X Dose B of ALXN2050 tablet under fasted conditions), Treatment B (single Dose A of ALXN2050 tablet under fasted conditions) and Treatment C (single Dose A of ALXN2050 tablet with a high-fat meal) on Day 1 of each treatment period. Washout period of at least 4 days between the ALXN2050 dose in each treatment period.
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C
- Treatment sequence ACB (Experimental): Participants will be administered Treatment A (3 X Dose B of ALXN2050 tablet under fasted conditions), Treatment C (single Dose A of ALXN2050 tablet with a high-fat meal) and Treatment B (single Dose A of ALXN2050 tablet under fasted conditions) on Day 1 of each treatment period. Washout period of at least 4 days between the ALXN2050 dose in each treatment period.
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C
- Treatment sequence BAC (Experimental): Participants will be administered Treatment B (single Dose A of ALXN2050 tablet under fasted conditions), Treatment A (3 X Dose B of ALXN2050 tablet under fasted conditions) and Treatment C (single Dose A of ALXN2050 tablet with a high-fat meal) and on Day 1 of each treatment period. Washout period of at least 4 days between the ALXN2050 dose in each treatment period.
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C
- Treatment sequence BCA (Experimental): Participants will be administered Treatment B (single Dose A of ALXN2050 tablet under fasted conditions), Treatment C (single Dose A of ALXN2050 tablet with a high-fat meal) and Treatment A (3 X Dose B of ALXN2050 tablet under fasted conditions) and on Day 1 of each treatment period. Washout period of at least 4 days between the ALXN2050 dose in each treatment period.
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C
- Treatment sequence CAB (Experimental): Participants will be administered Treatment C (single Dose A of ALXN2050 tablet with a high-fat meal), Treatment A (3 X Dose B of ALXN2050 tablet under fasted conditions) and Treatment B (single Dose A of ALXN2050 tablet under fasted conditions) on Day 1 of each treatment period. Washout period of at least 4 days between the ALXN2050 dose in each treatment period.
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C
- Treatment sequence CBA (Experimental): Participants will be administered Treatment C (single Dose A of ALXN2050 tablet with a high-fat meal), Treatment B (single Dose A of ALXN2050 tablet under fasted conditions) and Treatment A (3 X Dose B of ALXN2050 tablet under fasted conditions) on Day 1 of each treatment period. Washout period of at least 4 days between the ALXN2050 dose in each treatment period.
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C

INTERVENTIONS:
Drug: Treatment A — Participants will receive single Dose A dose of ALXN2050 tablet (3 × Dose B) orally under fasted conditions.
  Other Names: ACH-0145228
Drug: Treatment B — Participant will receive single Dose A of ALXN2050 tablet (1 × Dose A) orally under fasted conditions.
  Other Names: ACH-0145228
Drug: Treatment C — Participants will receive single Dose A of ALXN2050 tablet (1 × Dose A) orally with a high-fat meal.
  Other Names: ACH-0145228

SUMMARY:
This study will assess the Bioequivalence between 180 mg and 60 mg ALXN2050 Tablets and the Effect of Food on ALXN2050 Pharmacokinetics.

DETAILED DESCRIPTION:
This is a single-center, open-label, randomized, 3-period crossover study.

Screening of participants will occur within 28 days prior to the first dose of study intervention.

The study will comprise of 3 Treatment Periods: Treatment period 1, Treatment period 2, Treatment period 3. There will be a washout period of at least 4 days between the ALXN2050 dose in each treatment period.

Participants will be enrolled and will be randomized 1:1:1:1:1:1 to receive one of 6 treatment sequences (ABC, ACB, BAC, BCA, CAB, CBA).

On the morning of Day 1 of each of the 3 periods, participants will receive one of the following treatments as per the randomization scheme.

* Treatment A: Dose B of ALXN2050 tablet under fasted conditions
* Treatment B: A single Dose A dose of ALXN2050 tablet under fasted conditions
* Treatment C: A single Dose A dose of ALXN2050 tablet with a high-fat meal

Duration of study conduct (screening to follow-up): approximately 47 days.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who are healthy as determined by medical evaluation with no clinically significant or relevant abnormalities as determined by medical history, physical examination, neurological examination, vital signs, 12-lead ECG, and screening clinical laboratory profiles (hematology, biochemistry, coagulation, and urinalysis), that are reasonably likely to interfere with participation in or ability to complete the study, or to potentially confound interpretation of study results, as assessed by the Investigator or designee and Alexion Medical Monitor.
2. QT interval corrected using Fridericia's formula (QTcF) < 450 msec; QRS interval ≤ 110 msec; if > 110 msec, result will be confirmed by a manual over read; PR interval > 120 msec and < 220 msec at Screening
3. Body mass index (BMI) within the range 18.0 to 32.0 kg/m2, inclusive, with a minimum body weight of 50.0 kg at Screening.
4. Female participant of childbearing potential and male participants must follow protocol-specified contraception guidance.

Exclusion Criteria:

1. History of any medical (eg, cardiac, pulmonary, renal, or oncologic) or psychiatric condition or disease that, in the opinion of the Investigator or designee, might limit the participant's ability to complete or participate in this clinical study, confound the results of the study, or pose an additional risk to the participant by their participation in the study.
2. History of meningococcal infection.
3. History of clinically significant hypersensitivity or idiosyncratic reaction to the study interventions or related compounds.
4. History of clinically significant hypersensitivity reactions to commonly used antibacterial agents, including beta lactams, penicillin, aminopenicillins, fluoroquinolones, cephalosporins, and carbapenems, which in the opinion of the Investigator would make it difficult to properly provide either empiric antibiotic therapy or treat an active infection.
5. History of significant multiple and/or severe allergies
6. History of seizures.
7. History of head injury, or head trauma requiring medical evaluation.
8. History of drug or alcohol abuse
9. Current tobacco users or smoker
10. Diseases or conditions known to interfere with the absorption, distribution, metabolism or excretion of drugs. Any previous procedure, including history of stomach or intestinal surgery or resection, transjugular intrahepatic portosystemic shunts, or surgical shunt, that could alter absorption or excretion of orally administered drugs. Appendectomy, cholecystectomy, and hernia repair will be allowed if they were not associated with complications.
11. Any major surgery within 8 weeks of Screening.
12. Donation of whole blood from 3 months prior to first dose of study intervention or of plasma from 30 days prior to the first dose of study intervention.
13. History of malignancy within 5 years prior of Screening, with the exception of nonmelanoma skin cancer or carcinoma in situ of the cervix that has been treated with no evidence of recurrence.
14. Evidence of human immunodeficiency virus (HIV antibody positive) infection at screening.

18. Evidence of hepatitis B (positive hepatitis surface antigen [HBsAg]) or positive core antibody (anti-HBc) with negative surface antibody [anti-HBs]) or hepatitis C viral infection (HCV antibody positive) at screening.

19. Female participants who have a positive pregnancy test. 20. Vital signs out of the normal range as determined by the Investigator including body temperature ≥ 38°C.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2022-10-13 (Actual); Primary Completion 2023-01-05 (Actual); Study Completion 2023-01-05 (Actual)

PRIMARY OUTCOMES:
Cmax (Maximum observed plasma (peak) concentration of the drug) | Day 1, 2, 3 and 4 (Treatment Period 1, 2, 3) (each treatment period is of 4 days)
  To compare the single-dose PK of ALXN2050 when administered as Dose A tablet versus Dose B tablets.
  To determine the effect of food on the single-dose PK of Dose A of ALXN2050 tablet.
AUCt (Area under the concentration time curve from time zero to the last quantifiable concentration) | Day 1, 2, 3 and 4 (Treatment Period 1, 2, 3) (each treatment period is of 4 days)
  To compare the single-dose PK of ALXN2050 when administered as Dose A tablet versus Dose B tablets.
  To determine the effect of food on the single-dose PK of Dose A of ALXN2050 tablet.
AUC∞ (Area under the concentration time curve from time zero extrapolated to infinity) | Day 1, 2, 3 and 4 (Treatment Period 1, 2, 3) (each treatment period is of 4 days)
  To compare the single-dose PK of ALXN2050 when administered as Dose A tablet versus Dose B tablets.
  To determine the effect of food on the single-dose PK of Dose A of ALXN2050 tablet.
Tmax (Time corresponding to occurrence of Cmax) | Day 1, 2, 3 and 4 (Treatment Period 1, 2, 3) (each treatment period is of 4 days)
  To compare the single-dose PK of ALXN2050 when administered as Dose A tablet versus Dose B tablets.
  To determine the effect of food on the single-dose PK of Dose A of ALXN2050 tablet.
tlag (Time prior to the first measurable (non zero) concentration) | Day 1, 2, 3 and 4 (Treatment Period 1, 2, 3) (each treatment period is of 4 days)
  To compare the single-dose PK of ALXN2050 when administered as Dose A tablet versus Dose B tablets.
  To determine the effect of food on the single-dose PK of Dose A of ALXN2050 tablet.
t½ (Apparent terminal elimination half-life) | Day 1, 2, 3 and 4 (Treatment Period 1, 2, 3) (each treatment period is of 4 days)
  To compare the single-dose PK of ALXN2050 when administered as Dose A tablet versus Dose B tablets.
  To determine the effect of food on the single-dose PK of Dose A of ALXN2050 tablet.
λz (Terminal elimination rate constant) | Day 1, 2, 3 and 4 (Treatment Period 1, 2, 3) (each treatment period is of 4 days)
  To compare the single-dose PK of ALXN2050 when administered as Dose A tablet versus Dose B tablets.
  To determine the effect of food on the single-dose PK of Dose A of ALXN2050 tablet.
CL/F (Apparent clearance) | Day 1, 2, 3 and 4 (Treatment Period 1, 2, 3) (each treatment period is of 4 days)
  To compare the single-dose PK of ALXN2050 when administered as Dose A tablet versus Dose B tablets.
  To determine the effect of food on the single-dose PK of Dose A of ALXN2050 tablet.
Vd/F (Apparent volume of distribution during terminal phase) | Day 1, 2, 3 and 4 (Treatment Period 1, 2, 3) (each treatment period is of 4 days)
  To compare the single-dose PK of ALXN2050 when administered as Dose A tablet versus Dose B tablets.
  To determine the effect of food on the single-dose PK of Dose A of ALXN2050 tablet.

SECONDARY OUTCOMES:
Number of participants with treatment emergent adverse events (TEAE) and treatment emergent serious adverse events (TESAE) | From Screening (Day - 28 to Day -1) to Follow-up visit ((7 ± 2 days after Final Dose)/EOS) (approximately 47 days)
  To assess the safety and tolerability of a single-dose of ALXN2050 when administered as Dose A tablet and Dose B tablets.
  To assess the safety and tolerability of a single-dose of Dose A ALXN2050 tablet when administered either with or without food.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Alexion has a public commitment to allow requests for access to study data and will be supplying a protocol, CSR, and plain language summaries.
Supporting Information: Study Protocol, CSR

REFERENCES:
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=ALXN2050-HV-112&attachmentIdentifier=c2638bba-03be-4c83-9b8c-2921900328c3&fileName=ALXN2050-HV-112_CSR_synopsis_redacted.pdf&versionIdentifier=